CLINICAL TRIAL: NCT01722318
Title: A Randomized, 12-Week, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Assess the Safety and Efficacy of Plecanatide in Patients With Irritable Bowel Syndrome With Constipation (IBS-C)
Brief Title: The Plecanatide Irritable Bowel Syndrome With Constipation Study (IBS-C)
Acronym: CIBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP304-20212
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Irritable Bowel Syndrome Characterized by Constipation
MeSH Terms: interventions — plecanatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Plecanatide 0.3mg (Active Comparator): Plecanatide 0.3mg, one tablet by mouth daily for 12 weeks
  Interventions: Drug: Plecanatide
- Plecanatide 1.0mg (Active Comparator): Plecanatide 1.0mg one tablet by mouth daily for 12 weeks
  Interventions: Drug: Plecanatide
- Plecanatide 3.0mg (Active Comparator): Plecanatide 3.0mg, one tablet by mouth daily for 12 weeks
  Interventions: Drug: Plecanatide
- Plecanatide 9.0mg (Active Comparator): Plecanatide 9.0mg, one tablet by mouth daily for 12 weeks
  Interventions: Drug: Plecanatide
- Placebo (Placebo Comparator): Placebo, one tablet by mouth daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Plecanatide
  Other Names: Trulance
  Arms: Plecanatide 0.3mg; Plecanatide 1.0mg; Plecanatide 3.0mg; Plecanatide 9.0mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, 12-week, double-blind, placebo-controlled, dose-ranging study in patients with IBS-C.

DETAILED DESCRIPTION:
This is a randomized, 12-week, double-blind, placebo-controlled, dose-ranging study in patients with IBS-C. Patients will undergo a Screening Period to determine eligibility. After completing a Screening Visit patients will undergo a 2-week Pre-Treatment assessment using the Interactive Voice Response System (IVRS) during which they will complete daily assessments of bowel movements (BMs), stool consistency (Bristol Stool Form Scale- BSFS), abdominal pain or abdominal discomfort and other symptoms associated with IBS-C. Data from the two-week IVRS Pre-treatment assessment are used to define the patient's baseline from which change will be determined. Patients who meet all entry criteria will be randomized to one of five treatment groups ( 0.3mg,1.0mg,3.0mg,9mg,or Placebo) on Day 1 of the Treatment Period. Patients will take an oral dose of study drug daily (QD) for 12 weeks and continue the daily IVRS diaries (BMs, abdominal pain, other symptoms). On Weeks 2, 4, 8, and 12, patients will return to the clinic to undergo safety and efficacy assessments. For 2 weeks after completing dosing, (i.e., Post-Treatment Period), patients will continue to complete daily IVRS diaries. Patients will then return to the clinical site for a final follow-up visit (End of Study Visit). The planned duration of participation in this study will be approximately 112 days from signing of informed consent through post-treatment or 145 days if 30 day washout of a prohibited concomitant medication or stabilization of a medical condition is required before Pre-Treatment (up to 148 days, with all windows considered).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-75, inclusive
* Body Mass Index = 18-35 kg/m2, inclusive
* Meets modified Rome III criteria for irritable bowel syndrome with constipation which includes abdominal pain or discomfort for at least 3 days/month in the last 3 months with symptom onset for at least 6 months.
* Less than 3 CSBMs and less than 6 SBMs per week during the last 3 months.
* Hard or lumpy stools ≥ 25 % of defecations
* Patient has average abdominal pain intensity scores ≥ 3 (scale 0-10)for the combined 2 week pre-treatment period
* Patient is willing to discontinue use of supplemental fiber, laxatives, prescription and nonprescription medications, herbal or dietary supplements intended to treat constipation during the screening, pre-treatment, treatment and 2-week post-treatment periods
* Willing to maintain a stable diet during the study.
* Patients with hemorrhoids and/or diverticulosis (NOT diverticulitis) CAN be entered into the study.

Exclusion Criteria:

* Loose stool (mushy) or watery stool in the absence of any laxative or prohibited medicine for > 25% of BMs during the 3 months prior to screening visit OR during the 14 day pre-treatment period
* Patient has diarrhea-predominant or mixed ( diarrhea and constipation cycling or diarrhea and normal cycling) IBS.
* Active peptic ulcer disease not adequately treated or not stable
* History of cathartic colon, laxative, enema abuse, or ischemic colitis.
* Fecal impaction within 3 months of screening
* Patient has had /has any: structural abnormality of the GI tract or gastric bypass surgery, pelvic floor dysfunction, pseudo-obstruction, active infectious gastritis, diverticulitis, anal fissures or any disease or condition that can affect GI motility or defecation or can be associated with abdominal pain
* Unexplained and clinically significant "alarm symptoms" including lower GI bleeding, iron-deficiency anemia, weight loss or systemic signs of infection or colitis.
* Major surgery within 60 days of screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip B Miner, MD, Principal Investigator — Oklahoma Foundation for Digestive Research
Locations (99):
- United States (99):
  - Cahaba Research, Birmingham, Alabama
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Arrowhead Family Health Center PC dba Arrowhead Health Centers, Glendale, Arizona
  - Advanced Research Associates, LLC, Glendale, Arizona
  - Elite Clinical Trials, LLC, Phoenix, Arizona
  - Genova Clinical Research, Inc., Tucson, Arizona
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Advanced Rx Clinical Research, Inc., Artesia, California
  - GW Research, Inc., Chula Vista, California
  - SC Clinical Research, Inc., Garden Grove, California
  - Grossmont Center for Clinical Research, La Mesa, California
  - Community Clinical Trials, Orange, California
  - Healthcare Partners Medical Group, Pasadena, California
  - Medical Center for Clinical Research, San Diego, California
  - Memorial Research Medical Clinic d/b/a Orange Country Research Center, Tustin, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Consultants for Clinical Research of South Florida, Boynton Beach, Florida
  - Medical Research Unlimited, LLC, Hialeah, Florida
  - Eastern Research, Inc, Hialeah, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Jupiter Research, Inc., Jupiter, Florida
  - MNH Surgical Center, Maitland, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Genoma Research Group, Inc., Miami, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - South Medical Research Group, Inc., Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - Urology Center of Florida, Pompano Beach, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Meridien Research, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Georgia Regents University, Augusta, Georgia
  - Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - CTL Research, Eagle, Idaho
  - Medex Healthcare Research, Inc, Chicago, Illinois
  - Rockford Gastroenterology Associates, Rockford, Illinois
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Research Integrity, LLC, Owensboro, Kentucky
  - Delta Research Partners, LLC, Bastrop, Louisiana
  - Gastroenterology Research of New Orleans, Hammond, Louisiana
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Women Under Study, LLC, New Orleans, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Novex Clinical Research, LLC, New Bedford, Massachusetts
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - IHA Chelsea Family & Internal Medicine, Chelsea, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Ridgeview Research, Chaska, Minnesota
  - Prism Research, Saint Paul, Minnesota
  - The Center for Clinical Trials, Biloxi, Mississippi
  - Gastrointestinal Associates, PA, Jackson, Mississippi
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Montana Health Research Institute, Inc., Billings, Montana
  - Internal Medical Associates of Grand Island, PC, Grand Island, Nebraska
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - St. Luke's Hospital, New York, New York
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - MediSpect Medical Research, LLC, Boone, North Carolina
  - Clinical Trials of North Carolina, LLC, Cary, North Carolina
  - Carolina Digestive Health Associates, Charlotte, North Carolina
  - On Site Clinical, LLC, Charlotte, North Carolina
  - Carolina Digestive Health Associates, Davidson, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - LeBauer Research Associates, P.A., Greensboro, North Carolina
  - Medoff Medical / Vital re:Search, Greensboro, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Hometown Urgent Care and Occupational Health, Columbus, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Consultants in Gastroenterology, Columbia, South Carolina
  - Southeast Medical Research, North Charleston, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Chattanooga Medical Research LLC, Chattanooga, Tennessee
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Franklin Gastroenterology, PLLC, Franklin, Tennessee
  - Memphis Gastroenterology Group, PC, Germantown, Tennessee
  - Associates in Gastroenterology, Hermitage, Tennessee
  - Austin Center for Clinical Research, Austin, Texas
  - DCT-AACT, LLC dba Discovery Clinical Trials, Austin, Texas
  - Texas Tech Medical Center, El Paso, Texas
  - Centex Studies, Inc., Houston, Texas
  - North Texas Family Medicine, Plano, Texas
  - Quality Research, Inc., San Antonio, Texas
  - Physician PrimeCare Research Institute, PLLC dba Health Texas Research Institute, San Antonio, Texas
  - Pioneer Research Solutions, Inc., Sugar Land, Texas
  - New River Valley Research Institute, Christiansburg, Virginia
  - Blue Ridge Medical Research/Gastroenterology Associates of Central Virginia, Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Enrollment number in the Protocol Section was changed from 350 to 428 participants to reflect the actual enrollment number.
Groups:
- Plecanatide 0.3mg: Plecanatide 0.3mg, one tablet by mouth daily for 12 weeks
  Plecanatide
- Plecanatide 1.0mg: Plecanatide 1.0mg one tablet by mouth daily for 12 weeks
  Plecanatide
- Plecanatide 3.0mg: Plecanatide 3.0mg, one tablet by mouth daily for 12 weeks
  Plecanatide
- Plecanatide 9.0mg: Plecanatide 9.0mg, one tablet by mouth daily for 12 weeks
  Plecanatide
- Placebo: Placebo, one tablet by mouth daily for 12 weeks
  Placebo
Period: Overall Study
Arm/Group | Plecanatide 0.3mg | Plecanatide 1.0mg | Plecanatide 3.0mg | Plecanatide 9.0mg | Placebo
Started | 86 | 85 | 86 | 85 | 86
Completed | 72 | 65 | 66 | 65 | 68
Not Completed | 14 | 20 | 20 | 20 | 18

BASELINE CHARACTERISTICS:
Population: The Randomized Population (428 patients) in Participant Flow differs from the mITT Population (423 patients) because 1 patient was randomized and not dosed, 1 patient was dosed but had no post-baseline efficacy assessments, and 3 duplicate patient records (2 patients who were seen at 2 sites and 1 patient who was seen at 3 sites)
Groups:
- Total: Total of all reporting groups
Arm/Group | Plecanatide 0.3mg | Plecanatide 1.0mg | Plecanatide 3.0mg | Plecanatide 9.0mg | Placebo | Total
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85 | 423
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (12.02) | 44.6 (12.58) | 47.2 (12.89) | 45.3 (12.00) | 45.4 (12.02) | 45.9 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 67 | 70 | 70 | 69 | 344
  Male | 16 | 16 | 16 | 15 | 16 | 79

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly CSBMs Frequency Over the 12-Week Treatment Period (mITT Population)
Description: The primary efficacy endpoint was the change from baseline in the weekly CSBM frequency (CSBMs per week minus CSBMs per week at baseline) over a 12-week Treatment Period. A Complete Spontaneous Bowel Movement (CSBM) is a Bowel Movement (BM) that occurs in the absence of laxative use within 24 hours of the BM and the patient reports a feeling of complete evacuation.
Time Frame: 12 weeks Treatment Period
Population: The Modified Intent-to-Treat (mITT) population included all randomized patients who received ≥ 1 dose of study drug and ≥ 1 post-baseline BM assessment was the primary analysis population analyzed for efficacy endpoints.
Measure: Least Squares Mean (Standard Error); unit: CSBMs per week
Arm/Group | Plecanatide 0.3mg | Plecanatide 1.0mg | Plecanatide 3.0mg | Plecanatide 9.0mg | Placebo
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85
CSBMs per week | 1.28 (0.260) | 2.12 (0.265) | 2.74 (0.260) | 2.44 (0.262) | 1.27 (0.260)

2. Secondary Outcome: Change From Baseline in Abdominal Pain Intensity Scores Over 12-Week Treatment Period (mITT Population)
Description: Abdominal Pain was assessed in the patient's daily response on a scale of 0 to 10 where 0 is did not experience the symptom at all and 10 is experienced the worst.
Time Frame: 12-Week Treatment Period
Population: The mITT population included all randomized patients who received at least 1 dose of study drug and who had at least 1 post-baseline Bowel Movement (BM) assessment was the primary analysis population for efficacy endpoints.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Plecanatide 0.3mg | Plecanatide 1.0mg | Plecanatide 3.0mg | Plecanatide 9.0mg | Placebo
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85
scores on a scale | -1.5 (0.20) | -1.5 (0.20) | -2.0 (0.20) | -1.8 (0.20) | -1.4 (0.20)

3. Secondary Outcome: Change From Baseline in Stool Consistency (BSFS) Over 12-Week Treatment Period (mITT Population)
Description: The stool consistency of each bowel movement (BM) was assessed by patients using the 7-point Bristol Stool Form Scale [BSFS] from 1 to 7.
  1. = separate hard lumps like nuts (difficult to pass)
  2. = sausage shaped but lumpy
  3. = like a sausage but with cracks on its surface
  4. = like a sausage or snake, smooth and soft
  5. = soft blobs with clear-cut edges (passed easily)
  6. = fluffy pieces with ragged edges, a mushy stool
  7. = watery, no solid pieces (entirely liquid)
Time Frame: 12-Week Treatment Period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Plecanatide 0.3mg | Plecanatide 1.0mg | Plecanatide 3.0mg | Plecanatide 9.0mg | Placebo
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85
scores on a scale | 1.63 (0.143) | 1.81 (0.144) | 2.49 (0.143) | 2.24 (0.145) | 1.01 (0.143)

4. Secondary Outcome: Change From Baseline in Straining Scores Over 12-Week Treatment Period (mITT Population)
Description: The severity of straining (Straining Score) was rated by the patients using a 11-point scale (0-10) where 0 = none and 10 = very severe
Time Frame: 12-Week Treatment Period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Plecanatide 0.3mg | Plecanatide 1.0mg | Plecanatide 3.0mg | Plecanatide 9.0mg | Placebo
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85
score on a scale | -1.7 (0.23) | -1.5 (0.23) | -2.2 (0.23) | -2.1 (0.24) | -1.3 (0.23)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: A total of 428 patients were randomized and received at least one dose of medication except for one patient in the 0.3 mg plecanatide group. Therefore, a total of 427 patients were included in the safety population for adverse events reporting.
Arm/Group | Plecanatide 0.3mg | Plecanatide 1.0mg | Plecanatide 3.0mg | Plecanatide 9.0mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/85 | 0/85 | 1/86 | 2/85 | 0/86
Other Adverse Events (participants affected / at risk) | 18/85 | 29/85 | 19/86 | 31/85 | 12/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plecanatide 0.3mg (N=85) | Plecanatide 1.0mg (N=85) | Plecanatide 3.0mg (N=86) | Plecanatide 9.0mg (N=85) | Placebo (N=86)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plecanatide 0.3mg (N=85) | Plecanatide 1.0mg (N=85) | Plecanatide 3.0mg (N=86) | Plecanatide 9.0mg (N=85) | Placebo (N=86)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 8 (8) | 8 (9) | 10 (12) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2) | 4 (4) | 5 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 5 (5) | 3 (5) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 5 (5) | 3 (3) | 8 (8) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes